CLINICAL TRIAL: NCT03326986
Title: A Single Ascending Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-7252 in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics Study of MK-7252 in Healthy Adult Participants (MK-7252-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7252-001; 2017-003407-22 (EudraCT Number); MK-7252-001 (Other: Merck)
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Pharmacokinetics; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Panel A (Experimental): Participants receive either a single dose of MK-7252 or Placebo in a fasted state in each of five alternating treatment dosing periods as indicated. The planned dose levels include: Placebo for MK-7252, 1 mg of MK-7252, 6 mg of MK-7252, 24 mg of MK-7252, 72 mg of MK-7252, and 108 mg of MK-7252. There is a minimum of a 7-day washout period between each treatment period or dose administration. The planned dose levels may be adjusted downward or replaced based on evaluation of safety, tolerability, pharmacokinetic and/or pharmacodynamic data observed after previous treatment periods
  Interventions: Drug: MK-7252; Drug: Placebo
- Panel B (Experimental): Participants receive either a single dose of MK-7252 or Placebo in a fasted state in each of five alternating treatment dosing periods as indicated. The planned dose levels include: Placebo for MK-7252, 3 mg of MK-7252, 12 mg of MK-7252, 48 mg of MK-7252, 72 mg of MK-7252, and 162 mg of MK-7252. There is a minimum of a 7-day washout period between each treatment period or dose administration. The planned dose levels may be adjusted downward or replaced based on evaluation of safety, tolerability, pharmacokinetic and/or pharmacodynamic data observed after previous treatment periods
  Interventions: Drug: MK-7252; Drug: Placebo
- Panel C (Experimental): Participants receive either a single dose of MK-7252 or Placebo in up to 5 treatment dosing periods as indicated: Placebo for MK-7252, 120 mg of MK-7252 in a fasted state, 240 mg of MK-7252, 360 mg of MK-7252, 540 mg of MK-7252, and 120 mg of MK-7252 in a fed state. There is a minimum of a 7-day washout period between each treatment period or dose administration. The planned dose levels may be adjusted downward or replaced based on evaluation of safety, tolerability, pharmacokinetic and/or pharmacodynamic data observed after previous treatment periods
  Interventions: Drug: MK-7252; Drug: Placebo

INTERVENTIONS:
Drug: MK-7252 — 1 mg/mL or 20 mg/mL of powder for oral suspension administered with a water volume that brings the total ingested volume to approximately 240 mL
Drug: Placebo — Placebo powder for oral suspension administered with a water volume that brings the total ingested volume to approximately 240 mL

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of MK-7252 in healthy adults. Participants receive ascending doses of MK-7252 over five treatment periods. Each treatment period is separated by a 7-day washout period.

Upon review of the interim safety and preliminary PK data of human exposure to date, Protocol Amendment 3 includes a third panel of participants, Panel C, to assess the PK of higher doses of MK-7252 and to assess the food effect of MK-7252.

DETAILED DESCRIPTION:
Three panels (Panels A, B, and C) of 8 healthy participants (n=6 MK-7252, n=2 placebo) are enrolled. In Panels A and B, participants will alternately receive single rising doses of MK-7252 or placebo for 5 treatment periods. In Panel C, participants will receive single rising doses of MK-7252 or placebo for up to 5 treatment periods. All doses in Panels A and B will be administered in the fasted state during the 5 treatment periods. Doses in Panel C will be administered in a fasted state in treatment periods 1 through 4 and the treatment period 1 dose will be repeated in a fed state during treatment period 5. Panel A will begin first. At least 3 days will elapse before participants in Panel B will receive the next higher dose. For all panels, there will be at least 7 days washout between treatment periods for any given participant. Participants may only be enrolled in one panel of the study. The planned dose levels may be adjusted downward or replaced based on evaluation of safety, tolerability, pharmacokinetic and/or pharmacodynamic data observed after previous treatment periods. All participants in the treatment periods of all panels (with exception of 120 mg fasted/fed periods in Panel C) will be randomly assigned to either study drug or placebo; that is a participant could be assigned to receive study drug in one period and placebo in another. As per the protocol allocation plan, the same participants in Panel C will receive 120 mg MK-7252 in a fasted and fed state. In addition, during any of the treatment periods if a participant demonstrates change in any one of the protocol-defined parameters lasting ≥2 hours, dose escalation in that participant will be halted and the participant may be withdrawn from the study or re-challenged at same dose or at a lower or divided dose. Participants that meet criteria listed will be followed up until parameters no longer meet stopping rule criteria.

During the study, participants in Panel A were planned to receive placebo, 1 mg, 6 mg, 24 mg, 72 mg and 108 mg, all in a fasted state in 5 periods. Participants in Panel B were planned to receive placebo, 3 mg, 12 mg, 48 mg, 72 mg and 162 mg, all in a fasted state in 5 periods. All periods in Panels A and B were conducted. Participants in Panel C were planned to receive placebo fasted, placebo fed, 120 mg fasted, 240 mg fasted, 360 mg fasted, 540 mg fasted, and 120 mg fed in 5 periods. Periods 4 and 5 were not conducted and, as a result, the 240 mg fasted, 360 mg fasted, 540 mg fasted, 120 mg fed, and placebo fed doses were not administered. A 180 mg fasted dose was added during Period 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of non-childbearing potential (Note: If postmenopausal female: participant is without menses for at least 1 year and has a documented follicle stimulating hormone [FSH] level in the postmenopausal range at pre-trial [screening] - OR - If surgically sterile female: participant is status post hysterectomy, oophorectomy or tubal ligation.)
* Body Mass Index (BMI) between 18.5 and 32 kg/m^2, inclusive. BMI = weight (kg)/height (m)^2.
* While in semi-recumbent position, has a systolic blood pressure ≤140 mmHg and diastolic blood pressure ≤90 mm Hg and a respiratory rate ≤20 breaths/min at the pre-study (screening) visit and prior to randomization.
* Judged to be in good health based on medical history, physical examination, vital sign measurements and electrocardiogram (ECG) performed prior to randomization.
* Non-smoker and/or has not used nicotine or nicotine-containing products (e.g., nicotine patch) for at least approximately 3 months.

Exclusion Criteria:

* Mentally or legally incapacitated, has significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years.
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* History of liver disease (chronic hepatitis, cirrhosis, etc.).
* History of cancer (malignancy). Exceptions include adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix and other malignancies which have been successfully treated ≥10 years prior to the pre-study (screening) visit.
* History of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Tests positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pre-study (screening) visit.
* Participated in another investigational study within 4 weeks (or 5 half-lives), whichever is greater, prior to the pre-study (screening) visit.
* QTc interval ≥470 msec (for males) and ≥480 msec (for females).
* Taken a Proton Pump Inhibitor (PPI) during the 5 days prior to start of study treatment.
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the post-study visit.
* Consumes >3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day.
* Consumes excessive amounts, defined as >6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day.
* Regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year. Participants must have a negative result for urine drug screen test prior to randomization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Universitair Ziekenhuis Gent ( Site 0001), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in Panels A and B received a single-rising dose of MK-7252 or placebo in 5 alternating dosing periods. Participants in Panel C received a single-rising dose of MK-7252 or placebo in 3/5 planned periods (P). A 180 mg dose was added (P3). P4-5 were not run so the 240, 360, 540, and 120 mg fed and placebo fed doses were not given.
Groups:
- Panel A: Within each of the 5 rising dose treatment periods, 6 participants received a single dose of MK-7252 (1 mg, 6 mg, 24 mg, 72 mg, or 108 mg) and 2 participants received placebo in a fasted state. Dosing periods alternated with Panel B.
- Panel B: Within each of the 5 rising dose treatment periods, 6 participants received a single dose of MK-7252 (3 mg, 12 mg, 48 mg, 72 mg, or 162 mg) and 2 participants received placebo in a fasted state. Dosing periods alternated with Panel A.
- Panel C: Within each of 3 single dose treatment periods, 6 participants received a single dose of MK-7252 (120 mg or 180 mg) and 2 participants received placebo in a fasted state. The 120 mg dose of MK-7252 was administered in the first 2 periods and the 180 mg dose was administered in the third period.
Period: Overall Study
Arm/Group | Panel A | Panel B | Panel C
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A | Panel B | Panel C | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (10.2) | 35.0 (9.5) | 34.4 (9.3) | 34.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 7 | 6 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have had a causal relationship with this treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. Adverse events are reported by dose taken at time of event and not by panel or period. The adverse events for placebo are pooled over periods across panels. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 21 weeks
Population: All participants who received at least 1 dose of study treatment and experienced an AE during the study period
Measure: Count of Participants; unit: Participants
Groups:
- MK-7252 1 mg: Single oral dose of 1 mg MK-7252 administered in a fasted state
- MK-7252 3 mg: Single oral dose of 3 mg MK-7252 administered in a fasted state
- MK-7252 6 mg: Single oral dose of 6 mg MK-7252 administered in a fasted state
- MK-7252 12 mg: Single oral dose of 12 mg MK-7252 administered in a fasted state
- MK-7252 24 mg: Single oral dose of 24 mg MK-7252 administered in a fasted state
- MK-7252 48 mg: Single oral dose of 48 mg MK-7252 administered in a fasted state
- MK-7252 72 mg: Single oral dose of 72 mg MK-7252 administered in a fasted state
- MK-7252 108 mg: Single oral dose of 108 mg MK-7252 administered in a fasted state
- MK-7252 120 mg: Single oral dose of 120 mg MK-7252 administered in a fasted state
- MK-7252 162 mg: Single oral dose of 162 mg MK-7252 administered in a fasted state
- MK-7252 180 mg: Single oral dose of 180 mg MK-7252 administered in a fasted state
- Placebo: Single oral dose of placebo to match MK-7252 administered in a fasted state
Arm/Group | MK-7252 1 mg | MK-7252 3 mg | MK-7252 6 mg | MK-7252 12 mg | MK-7252 24 mg | MK-7252 48 mg | MK-7252 72 mg | MK-7252 108 mg | MK-7252 120 mg | MK-7252 162 mg | MK-7252 180 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 8 | 6 | 5 | 22
Participants | 2 | 5 | 4 | 5 | 5 | 4 | 7 | 5 | 6 | 4 | 2 | 15

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have had a causal relationship with this treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. Discontinuations are reported by dose taken at time of event. The discontinuations for placebo are pooled over periods across panels. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 19 weeks
Population: All participants who received at least 1 dose of study treatment and discontinued during the study period
Measure: Count of Participants; unit: Participants
Arm/Group | MK-7252 1 mg | MK-7252 3 mg | MK-7252 6 mg | MK-7252 12 mg | MK-7252 24 mg | MK-7252 48 mg | MK-7252 72 mg | MK-7252 108 mg | MK-7252 120 mg | MK-7252 162 mg | MK-7252 180 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 8 | 6 | 5 | 22
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

3. Secondary Outcome: MK-7252 Area Under the Concentration-Time Curve From Zero to Infinity (AUC0-∞)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 AUC0-∞ reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. Pharmacokinetic (PK) results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma AUC0-∞ following a high-fat breakfast (fed state) was planned to be compared to the plasma AUC0-∞ in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1) and 0.25, 0.5, 1, 2, 4, 8, 10, 12, 24, 48, and 72 hours postdose
Population: All participants who received study treatment and complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint. Periods (P) 4-5 of Panel C were not conducted; the planned 120 mg fed dose (P 5) was not administered.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr•nmol/L
Groups:
- Panel A MK-7252 1 mg: Single oral dose of 1 mg MK-7252 administered in a fasted state
- Panel B MK-7252 3 mg: Single oral dose of 3 mg MK-7252 administered in a fasted state
- Panel A MK-7252 6 mg: Single oral dose of 6 mg MK-7252 administered in a fasted state
- Panel B MK-7252 12 mg: Single oral dose of 12 mg MK-7252 administered in a fasted state
- Panel A MK-7252 24 mg: Single oral dose of 24 mg MK-7252 administered in a fasted state
- Panel B MK-7252 48 mg: Single oral dose of 48 mg MK-7252 administered in a fasted state
- Panel A MK-7252 72 mg: Single oral dose of 72 mg MK-7252 administered in Panel A in a fasted state
- Panel B MK-7252 72 mg: Single oral dose of 72 mg MK-7252 administered Panel B in a fasted state
- Panel A MK-7252 108 mg: Single oral dose of 108 mg MK-7252 administered in a fasted state
- Panel B MK-7252 162 mg: Single oral dose of 162 mg MK-7252 administered in a fasted state
- Panel C MK-7252 120 mg Period 1: Single oral dose of 120 mg MK-7252 administered in Panel C Period 1 in a fasted state
- Panel C MK-7252 120 mg Period 2: Single oral dose of 120 mg MK-7252 administered in Panel C Period 2 in a fasted state
- Panel C MK-7252 180 mg Period 3: Single oral dose of 180 mg MK-7252 administered in Panel C Period 3 in a fasted state
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr•nmol/L | NA [NA to NA] — Geometric mean and 95% confidence interval were not calculated for the 1 mg dose: there were insufficient data points above the lower limit of quantification of the assay (2.74 nM) to calculate the AUC0-∞ at this dose level. | NA [NA to NA] — Geometric mean and 95% confidence interval were not calculated for the 3 mg dose: there were insufficient data points above the lower limit of quantification of the assay (2.74 nM) to calculate the AUC0-∞ at this dose level. | 288 [195 to 427] | 583 [394 to 862] | 1190 [805 to 1750] | 2040 [1390 to 3000] | 5090 [3460 to 7490] | 3500 [2380 to 5160] | 6680 [4530 to 9840] | 9840 [6690 to 14500] | 7260 [4930 to 10700] | 5520 [3720 to 8170] | 10300 [6970 to 15300]

4. Secondary Outcome: MK-7252 Area Under the Concentration-Time Curve From Zero to 24 Hours Postdose (AUC0-24hr)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 AUC0-24hr reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma AUC0-24hr following a high-fat breakfast (fed state) was planned to be compared to the plasma AUC0-24hr in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, 12, and 24 hours postdose
Population: All participants who received study treatment and complied with the protocol sufficiently to ensure that data were likely to exhibit the effects of the treatment, according to the underlying scientific model and had data available for endpoint. Periods (P) 4 and 5 of Panel C were not conducted; the planned 120 mg fed dose (P5) was not administered.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr•nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr•nmol/L | 47.8 [32.4 to 70.4] | 122 [82.4 to 179] | 279 [189 to 411] | 559 [379 to 824] | 1150 [781 to 1700] | 2030 [1380 to 3000] | 5210 [3530 to 7680] | 3490 [2370 to 5150] | 6420 [4350 to 9470] | 9530 [6460 to 14100] | 7240 [4900 to 10700] | 5510 [3710 to 8200] | 10300 [6910 to 15300]

5. Secondary Outcome: MK-7252 Area Under the Concentration-Time Curve From Zero to 12 Hours Postdose (AUC0-12hr)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 AUC0-12hr reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma AUC0-12hr following a high-fat breakfast (fed state) was planned to be compared to the plasma AUC0-12hr in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, and 12 hours postdose
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr•nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr•nmol/L | 47.8 [32.5 to 70.4] | 121 [82.5 to 179] | 278 [189 to 409] | 558 [379 to 822] | 1140 [775 to 1680] | 2020 [1370 to 2980] | 5130 [3480 to 7540] | 3450 [2340 to 5070] | 6220 [4220 to 9160] | 9240 [6270 to 13600] | 7170 [4860 to 10600] | 5480 [3690 to 8130] | 10200 [6840 to 15100]

6. Secondary Outcome: MK-7252 Area Under the Concentration-Time Curve From Zero to Last Measurable Concentration (AUClast)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 AUClast reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma AUClast following a high-fat breakfast (fed state) was planned to be compared to the plasma AUClast in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, 12, 24, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: hr•nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr•nmol/L | 38.7 [26.0 to 57.6] | 101 [68.1 to 151] | 250 [168 to 371] | 543 [365 to 808] | 1130 [757 to 1680] | 2030 [1360 to 3020] | 5170 [3470 to 7690] | 3420 [2300 to 5090] | 6330 [4250 to 9420] | 9750 [6550 to 14500] | 7250 [4860 to 10800] | 5500 [3670 to 8260] | 10300 [6860 to 15500]

7. Secondary Outcome: MK-7252 Maximal Plasma Concentration (Cmax)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 Cmax reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma Cmax following a high-fat breakfast (fed state) was planned to be compared to the plasma Cmax in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, 12, 24, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol/L | 21.2 [15.4 to 29.4] | 51.7 [37.4 to 71.5] | 117 [84.6 to 162] | 220 [159 to 305] | 447 [323 to 618] | 830 [600 to 1150] | 1860 [1340 to 2570] | 1380 [997 to 1910] | 2290 [1660 to 3170] | 3380 [2440 to 4670] | 3160 [2280 to 4380] | 2550 [1820 to 3580] | 3880 [2760 to 5440]

8. Secondary Outcome: MK-7252 Plasma Concentration at 12 Hours Postdose (C12hr)
Description: Blood samples were obtained 12 hours postdose to calculate the plasma MK-7252 C12hr reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. For participants in a given dose that had C12hr values less than the lower limit of quantification (LLOQ), the C12hr value was imputed as half x LLOQ. The LLOQ was 2.74 nmol/L. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma C12hr following a high-fat breakfast (fed state) was planned to be compared to the plasma C12hr in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: 12 hours postdose
Population: as for outcome 4
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol/L | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C12hr values for the 1 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C12hr values for the 3 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C12hr values for the 6 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C12hr values for the 12 mg dose level being below the LLOQ (2.74 nmol/L). | 2.19 [1.17 to 4.10] | 2.95 [1.57 to 5.51] | 11.7 [6.29 to 21.7] | 7.06 [3.80 to 13.1] | 21.0 [11.2 to 39.2] | 31.8 [17.0 to 59.6] | 10.4 [5.59 to 19.3] | 7.16 [3.76 to 13.7] | 16.7 [8.77 to 31.9]

9. Secondary Outcome: MK-7252 Plasma Concentration at 24 Hours Postdose (C24hr)
Description: Blood samples were obtained 24 hours postdose to calculate the plasma MK-7252 C24hr reported as back-transformed least squares mean and confidence interval calculated using a linear mixed effects model performed on natural log-transformed values. For participants in a given dose that had C24hr values less than the lower limit of quantification (LLOQ), the C24hr value was imputed as half x LLOQ. The LLOQ was 2.74 nmol/L. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma C24hr following a high-fat breakfast (fed state) was planned to be compared to the plasma C24hr in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: 24 hours postdose
Population: All participants who received study treatment, complied with the protocol to ensure data were likely to exhibit effects of treatment according to the scientific model, and had data available for endpoint. Periods 4-5 of Panel C was not conducted and planned 120 mg fed dose not administered. Analysis was not performed due to values being <LLOQ.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
nmol/L | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 1 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 3 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 6 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 12 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 24 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 48 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 72 mg dose in level in Panel A being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 72 mg dose level in Panel B being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 108 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 162 mg dose level being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 120 mg dose level in Panel C Period 1 being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 120 mg dose level in Panel C Period 2 being below the LLOQ (2.74 nmol/L). | NA [NA to NA] — Geometric least squares mean and 90% confidence interval were not calculated due to C24hr values for the 180 mg dose level in Panel C Period 3 being below the LLOQ (2.74 nmol/L).

10. Secondary Outcome: MK-7252 Time to Reach Maximal Concentration (Tmax)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 Tmax. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma Tmax following a high-fat breakfast (fed state) was planned to be compared to the plasma Tmax in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, 12, 24, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr | 1.00 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 1.00]

11. Secondary Outcome: MK-7252 Apparent Terminal Half-life (t½)
Description: Blood samples were obtained predose (Day 1) and at designated times postdose to calculate the plasma MK-7252 t½ reported as Geometric Mean with Percent Geometric Coefficient of Variation. PK results were reported by dose taken in Panels A and B. For Panel C, PK results were reported by dose taken and by individual period. Periods in a panel were not conducted if it became evident that exposures at the escalated dosing would not adequately reach the projected PK target. Although the plasma t½ following a high-fat breakfast (fed state) was planned to be compared to the plasma t½ in the fasted stated in Panel C, the fed state dose was not administered.
Time Frame: Predose (Day 1), 0.25, 0.5, 1, 2, 4, 8, 10, 12, 24, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
hr | NA (NA) — Geometric mean and 95% confidence interval were not calculated for the 1 mg dose: there were insufficient data points above the lower limit of quantification of the assay (2.74 nM) to calculate the t½ at this dose level. | NA (NA) — Geometric mean and 95% confidence interval were not calculated for the 3 mg dose: there were insufficient data points above the lower limit of quantification of the assay (2.74 nM) to calculate the t½ at this dose level. | 1.29 (12.18) | 1.34 (14.99) | 1.60 (19.86) | 1.35 (9.93) | 1.76 (60.34) | 1.59 (19.54) | 3.09 (81.14) | 5.97 (92.18) | 1.96 (52.80) | 2.40 (71.03) | 2.90 (152.97)

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 4 Hours
Description: Assessment of the change from baseline in SBP was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 SBP measurements: baseline and 4 hours postdose. SBP results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in SBP and a negative number indicates a decrease in SBP.
Time Frame: Baseline (Predose Day 1) and 4 hours postdose
Population: All participants who received at least 1 dose of study treatment and had SBP assessments at baseline and 4 hours postdose
Measure: Mean (Standard Error); unit: mmHg
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
mmHg | 5.61 (1.94) | 1.56 (2.57) | 0.50 (2.66) | 4.39 (2.08) | 6.78 (3.71) | 12.17 (1.57) | 14.00 (4.28) | 9.83 (0.84) | 11.28 (1.90) | 5.33 (2.15) | 18.17 (7.65) | 3.80 (4.15) | 6.13 (4.52) | 3.22 (1.84)

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 24 Hours
Description: Assessment of the change from baseline in SBP was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 SBP measurements: baseline and 24 hours postdose. SBP results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in SBP and a negative number indicates a decrease in SBP.
Time Frame: Baseline (Predose Day 1) and 24 hours postdose
Population: All participants who received at least 1 dose of study treatment and had SBP assessments at baseline and 24 hours postdose
Measure: Mean (Standard Error); unit: mmHg
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
mmHg | 2.83 (3.40) | 0.89 (3.00) | -1.11 (1.56) | -3.56 (2.47) | -0.17 (2.75) | -0.56 (2.48) | 7.56 (1.32) | 3.56 (1.81) | 0.22 (3.36) | 3.17 (1.61) | 4.67 (3.51) | -0.13 (4.98) | 7.27 (3.86) | 5.84 (1.48)

14. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at 4 Hours
Description: Assessment of the change from baseline in DBP was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 DBP measurements: baseline and 4 hours postdose. DBP results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in DBP and a negative number indicates a decrease in DBP.
Time Frame: Baseline (Predose Day 1) and 4 hours postdose
Population: All participants who received at least 1 dose of study treatment and had DBP assessments at baseline and 4 hours postdose
Measure: Mean (Standard Error); unit: mmHg
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
mmHg | 1.11 (1.77) | 1.61 (1.06) | 0.33 (1.88) | 2.28 (3.24) | 6.33 (1.55) | 6.22 (1.56) | 5.50 (2.03) | 7.28 (2.24) | 4.61 (1.24) | 5.33 (1.43) | 5.28 (1.24) | 11.27 (3.12) | 5.67 (1.96) | 0.61 (0.83)

15. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at 24 Hours
Description: Assessment of the change from baseline in DBP was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 DBP measurements: baseline and 24 hours postdose. DBP results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in DBP and a negative number indicates a decrease in DBP.
Time Frame: Baseline (Predose Day 1) and 24 hours postdose
Population: All participants who received at least 1 dose of study treatment and had DBP assessments at baseline and 24 hours postdose
Measure: Mean (Standard Error); unit: mmHg
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
mmHg | 0.61 (1.31) | 2.78 (3.13) | -2.67 (2.86) | -3.33 (2.23) | 2.33 (1.69) | -1.11 (2.03) | 2.11 (1.91) | 1.72 (1.62) | -0.78 (2.49) | 4.11 (1.89) | 1.28 (1.59) | 4.00 (1.15) | 4.73 (1.16) | 1.99 (0.83)

16. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 4 Hours
Description: Assessment of the change from baseline in HR was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 HR measurements: baseline and 4 hours postdose. HR results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in HR and a negative number indicates a decrease in HR.
Time Frame: Baseline (Predose Day 1) and 4 hours postdose
Population: All participants who received at least 1 dose of study treatment and had HR assessments at baseline and 4 hours postdose
Measure: Mean (Standard Error); unit: beats per minute
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
beats per minute | -4.22 (1.82) | -0.28 (2.66) | -1.22 (1.68) | -0.89 (1.76) | 0.22 (0.88) | 0.17 (1.72) | 6.83 (7.05) | 2.28 (2.99) | 0.83 (2.21) | 1.33 (2.10) | 2.17 (6.07) | -1.53 (1.36) | 1.27 (2.15) | -1.27 (0.91)

17. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 24 Hours
Description: Assessment of the change from baseline in HR was obtained using a validated, semi-automated oscillometric device. Baseline was defined as the average of predose measurements. A measurement set was considered 2 HR measurements: baseline and 24 hours postdose. HR results are reported by dose taken. Placebo measurements are pooled over periods across panels. A positive number indicates an increase in HR and a negative number indicates a decrease in HR.
Time Frame: Baseline (Predose Day 1) and 24 hours postdose
Population: All participants who received at least 1 dose of study treatment and had HR assessments at baseline and 24 hours postdose
Measure: Mean (Standard Error); unit: beats per minute
Units Other Than Participants: Measurement sets
Arm/Group | Panel A MK-7252 1 mg | Panel B MK-7252 3 mg | Panel A MK-7252 6 mg | Panel B MK-7252 12 mg | Panel A MK-7252 24 mg | Panel B MK-7252 48 mg | Panel A MK-7252 72 mg | Panel B MK-7252 72 mg | Panel A MK-7252 108 mg | Panel B MK-7252 162 mg | Panel C MK-7252 120 mg Period 1 | Panel C MK-7252 120 mg Period 2 | Panel C MK-7252 180 mg Period 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 22
Number analyzed (Measurement sets) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 25
beats per minute | -2.78 (2.01) | 2.72 (2.03) | 1.83 (1.38) | 3.89 (1.55) | 2.89 (1.19) | 1.67 (1.41) | 2.94 (1.73) | 2.17 (2.15) | -0.61 (1.46) | 2.67 (2.18) | -0.72 (2.53) | 1.40 (1.26) | 2.33 (1.13) | 2.23 (1.27)

ADVERSE EVENTS:
Time Frame: Up to approximately 21 weeks
Description: The safety population includes all participants who received at least 1 dose of study treatment. Adverse events are reported by dose taken at time of event and not by panel or period. Post-study adverse events were pooled across all arms in the study (MK-7252 and placebo).
Groups:
- MK-7252 72 mg: Single oral dose of 72 mg of MK-7252 administered in a fasted state
- MK-7252 120 mg: Single oral dose of 120 mg of MK-7252 administered in a fasted state
- MK-7252 180 mg: Single oral dose of 180 mg of MK-7252 administered in a fasted state
- Post-Study: MK-7252 or placebo as a single dose in the post-study period administered in a fasted state
Arm/Group | MK-7252 1 mg | MK-7252 3 mg | MK-7252 6 mg | MK-7252 12 mg | MK-7252 24 mg | MK-7252 48 mg | MK-7252 72 mg | MK-7252 108 mg | MK-7252 120 mg | MK-7252 162 mg | MK-7252 180 mg | Placebo | Post-Study
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/8 | 0/6 | 0/5 | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/8 | 0/6 | 0/5 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 2/6 | 5/6 | 4/6 | 5/6 | 5/6 | 4/6 | 7/12 | 5/6 | 6/8 | 4/6 | 2/5 | 15/22 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MK-7252 1 mg (N=6) | MK-7252 3 mg (N=6) | MK-7252 6 mg (N=6) | MK-7252 12 mg (N=6) | MK-7252 24 mg (N=6) | MK-7252 48 mg (N=6) | MK-7252 72 mg (N=12) | MK-7252 108 mg (N=6) | MK-7252 120 mg (N=8) | MK-7252 162 mg (N=6) | MK-7252 180 mg (N=5) | Placebo (N=22) | Post-Study (N=24)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 8 (8) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/86/NCT03326986/Prot_SAP_000.pdf